CLINICAL TRIAL: NCT01689012
Title: A Pilot Study of the Efficacy of a Facial Exercise Program
Brief Title: The Effect of Facial Exercise on the Appearance of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STU68255
Record Dates: First submitted 2012-09-14; First posted 2012-09-20 (Estimated); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Facial Exercise (Experimental)
  Interventions: Behavioral: Facial Exercise

INTERVENTIONS:
Behavioral: Facial Exercise

SUMMARY:
This study seeks to evaluate the effects of facial exercises on aging of the face.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-65 years
* No significant medical illness
* No chronic smokers
* Subject with mild to moderate facial atrophy
* Subjects who provide and interest and who understand the importance of consistently executing the program daily.
* Subjects with the willingness and ability to understand and provide informed consent.

Exclusion Criteria:

* Under 40 years of age, Over 65 years of age
* Pregnant or lactating
* Subjects who have ever had any invasive cosmetic procedure, including facelifts, neck lifts, laser resurfacing, dermabrasion, or liposuction
* Subjects who have non-invasive or minimally invasive cosmetic procedures, such a non-ablative lasers, medium-depth or deeper chemical peels, injectable neurotoxins or fillers, within the past year.
* Subjects who have used topical or oral retinoids within the past year.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Improvement of face and neck after facial exercise compared to baseline | up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States